CLINICAL TRIAL: NCT01258374
Title: Dual Therapy With Raltegravir 400 mg BID and Darunavir/Ritonavir 800/100 mg QD in HIV Infected Patients Failing to Nucleoside Reverse Transcriptase Inhibitors Based Regimens
Brief Title: Dual Therapy With Raltegravir and Darunavir/Ritonavir in HIV Infected Patients.
Acronym: RALDAR
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Mallolas Masferrer, MD, PhD, Hospital Clinic of Barcelona
Other Study IDs: RALDAR-HCB
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-08

CONDITIONS: Integrase Inhibitors, HIV; HIV PROTEASE INHIB
Keywords: Pharmacokinetics, raltegravir, darunavir, NRTI sparing regimen
MeSH Terms: interventions — Raltegravir Potassium; Darunavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm with dual therapy: Dual therapy RAL 400 mg bid + DRV/r 800/100 mg QD
  Interventions: Drug: Raltegravir; Drug: Darunavir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir, 400 mg bid
  Other Names: Isentress
Drug: Darunavir — Darunavir, 800 mg QD + ritonavir 100 mg QD
  Other Names: Prezista, Norvir.

SUMMARY:
While 3-drug regimens remain standard of care, concerns exist regarding the safety of multi-drug regimens taken for a lifetime. Problems with nucleoside analogue therapy prompted successful trials with ritonavir (RTV) boosted PI monotherapy, however long term safety and efficacy of such regimens remains unknown. Clinical trials have shown Raltegravir (RAL) to have potent activity when patients have few active background drugs; it has a superior lipid profile compared with EFV and LPV/RTV. Darunavir/r (DRV) is a potent, well tolerated PI with few GI side effects and lipid disturbances and with a high genetic barrier. The investigators hypothesized that RAL/DRV would be a well tolerated and effective regimen for those patients who are failing nucleoside reverse transcriptase inhibitors based regimens, due to poor tolerability or resistance. The investigators also would like to explore the plasma pharmacokinetics of Raltegravir combined with Darunavir in a sub-group of 12 HIV-infected patients.

DETAILED DESCRIPTION:
Hypothesis

* NRTI-sparing regimens are attractive options to avoid NRTI-associated toxicity and to provide a full active regimen in patients with some extent of NRTI resistance.
* Raltegravir (RAL) and Darunavir (DRV) are potent "third drugs" and they provide a synergistic inhibition of 2 different steps in HIV replication.
* DRV has a high genetic barrier, and could be an excellent accompanying drug for Raltegravir, providing a potent, safe and well tolerated dual therapy to patients who are failing NNRTI based treatments.

Objectives:

* To describe the safety, tolerability and efficacy of the combination of Raltegravir and Darunavir after 24 weeks of follow up in HIV infected patients failing a NRTI based regimen.
* To describe plasma pharmacokinetics of Raltegravir when combined with Darunavir 800mg QD in HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Naïve to Raltegravir.
* CD4 cell count above 200 cell/mm3.
* No history of failure to PI containing regimens.
* No evidence of PI mutations (IAS-mutation list) by genotype test.
* Failing to a NRTI based regimen.
* The treating physician decides a NRTI sparing regimen which includes DRV/r 800/100 mg QD plus Raltegravir 400 mg BID.
* Signed informed consent form
* In opinion of the investigator, the patient should be considered clinically stable and could follow regular visits as scheduled per protocol.

Exclusion Criteria:

* Patients receiving drugs considered contraindicated to Raltegravir and DRV/r. Contraindicated drugs are: rifampin, fenitoin, phenobarbital in the case of raltegravir. Pravastatin, astemizole, sildenafil, are contraindicated in combination with DRV/r.
* Pregnancy
* Documented PI mutations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 HIV-infected patients failing NRTI based regimens will be included . At least 12 of these patients will undergo a complete pharmacokinetic study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Mallolas, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Rebollar M, Munoz A, Perez I, Hidalgo S, Brunet M, Laguno M, Gonzalez A, Calvo M, Lonca M, Blanco JL, Martinez E, Gatell JM, Mallolas J. Pharmacokinetic study of dual therapy with raltegravir 400 mg twice daily and Darunavir/Ritonavir 800/100 mg once daily in HIV-1-infected patients. Ther Drug Monit. 2013 Aug;35(4):552-6. doi: 10.1097/FTD.0b013e31828d50ef. PMID 23851911

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The treating physician chose an NRTI-sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily. 15 patients were screenend and all of them were included and finish the study
Period: Overall Study
Arm/Group | Single Arm With Dual Therapy
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm With Dual Therapy
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 44 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Spain | 15

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of C-Trough, of Raltegravir (RAL) at a Dose of 400 mg Twice a Day Plus Darunavir/Ritonavir (DRV/RTV) at a Dose of 800/100 mg Once a Day in HIV-1-infected Patients Were Mesured After 15 Days of Therapy.
Description: Geometric mean of C-Trough, of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy.The treating physician chose an NRTI-sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily. All patients were RAL and DRV naive and had no evidence of protease inhibitor mutations.
Time Frame: After at least 15 days on therapy, patients were admitted for a 24-hour PK study. The moorning dose of RAL adn DRV/r was administered in the clinic with. Blood samples were drawn immediatly before breakfast and 0.5, 1,2,3,4,6,8,12 and 24 hours afterward.
Population: HIV-1-infected patients, receiving a NRTI-based regimen, naive to RAL, with no evidence of PI mutations by genotype test, and signed informed consent forms. 15 patients ere screened and enrolled
Measure: Geometric Mean (Full Range); unit: ng/ml
Groups:
- Single Arm With Dual Therapy: Fifteen patients were screened and enrolled, and all of them completed the study procedures. The treating physician chose an NRTI-sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily.
  Inclusion criteria were HIV-1-infected patients, receiving a NRTI-based regimen, naive to RAL, with no evidence of PI mutations by genotype test, and signed informed consent forms. All doses of RAL were administered in the morning and evening, orally with food (light meal). Patients were admitted to the hospital in the morning on day 15 and stayed for 12 hours after the last administration of RAL. The morning dose of RAL and DRV/ RTV was administered in the clinic with a light breakfast (200 mL of whole milk and a ham and cheese sandwich), and blood samples were drawn immediately before breakfast and 0.5 1, 2, 3, 4, 6, 8, 12, and 24 hours afterward
Arm/Group | Single Arm With Dual Therapy
Number analyzed (Participants) | 15
ng/ml
  C trough Darunavir | 1330 [1110 to 1760]
  C trough Raltegravir | 40 [30 to 80]
  C trough Ritonavir | 90 [70 to 140]
Statistical Analysis 1: Comparison: Single Arm With Dual Therapy; Test type: Other; p < 0.01, Noncompartmental modeling techniques — The PK paramaters reported as geometric means, were calculated using noncompartmental modelinf techniques (WinNolin; Pharsight Corporation, Mountain View, CA); The pharmacokinetic parameters calculated for DRV, RTV and RAL were trough plasma concentration (C trough), defined as the concentration at 24 or 12 h after observed dose, the maximum observed plasma concentration (C max), the area under the plasma concentration-time curve from 0 to 24 H (AUC 0-24) or 0 to 12 h (AUC 0-12) and the elimination half-life (t1/2). AUC and t1/2 were calculated using non using noncompartmental modeling techniques (WinNolin; Pharsight Corporation, Mountain View, CA). All of these PK parameters are reported as geometric means

2. Primary Outcome: Geometric Mean of AUC, of Raltegravir (RAL) at a Dose of 400 mg Twice a Day Plus Darunavir/Ritonavir (DRV/RTV) at a Dose of 800/100 mg Once a Day in HIV-1-infected Patients Were Mesured After 15 Days of Therapy.
Description: Geometric mean of AUC0 of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy. The treating physician chose an NRTI-Geometric mean of C-Trough, of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy.sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily. All patients were RAL and DRV naive and had no evidence of protease inhibitor mutations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng.h/mL
Arm/Group | Single Arm With Dual Therapy
Number analyzed (Participants) | 15
ng.h/mL
  AUC Raltegravir | 3050 [2530 to 5180]
  AUC Darunavir | 68,730 [58,970 to 86,480]
  AUC Ritonavir | 5470 [4500 to 7420]

3. Primary Outcome: Geometric Mean of C-max, of Raltegravir (RAL) at a Dose of 400 mg Twice a Day Plus Darunavir/Ritonavir (DRV/RTV) at a Dose of 800/100 mg Once a Day in HIV-1-infected Patients Were Mesured After 15 Days of Therapy.
Description: Geometric mean of C-max of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy. The treating physician chose an NRTI-Geometric mean of C-max, of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy.sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily. All patients were RAL and DRV naive and had no evidence of protease inhibitor mutations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Single Arm With Dual Therapy
Number analyzed (Participants) | 15
ng/mL
  Cmax Darunavir | 7630 [6740 to 9000]
  Cmax Raltegravir | 970 [840 to 2270]
  Cmax Ritonavir | 490 [410 to 630]

4. Primary Outcome: Geometric Mean of t1/2, of Raltegravir (RAL) at a Dose of 400 mg Twice a Day Plus Darunavir/Ritonavir (DRV/RTV) at a Dose of 800/100 mg Once a Day in HIV-1-infected Patients Were Mesured After 15 Days of Therapy
Description: Geometric mean of t1/2 of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy. The treating physician chose an NRTI-Geometric mean of t1/2, of raltegravir (RAL) at a dose of 400 mg twice a day plus darunavir/ritonavir (DRV/RTV) at a dose of 800/100 mg once a day in HIV-1-infected patients were mesured after 15 days of therapy.sparing regimen because of toxicity or resistance mutations to NRTIs, which included DRV/RTV 800/100 mg once daily plus RAL 400 mg twice daily. All patients were RAL and DRV naive and had no evidence of protease inhibitor mutations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | Single Arm With Dual Therapy
Number analyzed (Participants) | 15
h
  t1/2 Darunavir | 10.91 [9.20 to 13.99]
  t1/2 Raltegravir | 2.68 [1.97 to 4.40]
  t1/2 Ritonavir | 9.48 [8.15 to 11.63]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Single Arm With Dual Therapy
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The main limitation of our study is that it is a single-arm PK study and, thus, the effect of the introduction or withdrawal of one drug over the other cannot be compared.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes